CLINICAL TRIAL: NCT01251809
Title: A Randomized, Multi-centre, Parallel-group, Open Label, Oncaspar® Controlled Dose Ranging Trial of Three Doses of Pegylated Recombinant Asparaginase in Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukaemia
Brief Title: Trial of Oncaspar® and Three Doses of Pegylated Recombinant Asparaginase in Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukaemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-PEGASP.1/adults
Record Dates: First submitted 2010-11-26; First posted 2010-12-02 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Acute Lymphoblastic Leukaemia
Keywords: Asparaginase; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PEG-rASNase 500 (Experimental): 500 U/m2 BSA at day 0
  Interventions: Drug: PEG-rASNase
- PEG-rASNase 1000 (Experimental): 1000 U/m2 BSA at day 0
  Interventions: Drug: PEG-rASNase
- PEG-rASNase 1500 (Experimental): 1500 U/m2 at day 0
  Interventions: Drug: PEG-rASNase
- Oncaspar (Active Comparator): 2000 U/m2 at day 0
  Interventions: Drug: Oncaspar

INTERVENTIONS:
Drug: Oncaspar — 2000 U/m2 BSA, single infusion
  Arms: Oncaspar
Drug: PEG-rASNase — 500, 1000 or 1500 U/m2 BSA single infusion
  Arms: PEG-rASNase 1000; PEG-rASNase 1500; PEG-rASNase 500

SUMMARY:
This is an assessment of efficacy and safety of three different doses of pegylated recombinant asparaginase (PEG-rASNase) in comparison to Oncaspar® during treatment of adults with de novo acute lymphoblastic leukaemia (ALL). This study will provide first data for determining specific asparaginase doses to yield various durations of L-asparagine (ASN) depletion which are required within different treatment phases of ALL therapy.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated acute lymphoblastic leukaemia (pro-B, common, pre-B, early T, thymic T, mature T)
* Age 18 years - 55 years
* Treatment according to German Multicenter Trials for adult Acute Lymphoblastic Leukaemia (GMALL) 07/2003 protocol or subsequent GMALL protocols for patients with de novo ALL
* Written informed consent
* Women of child-bearing potential or partner of men with child-bearing potential must use a highly effective method of contraception
* Negative pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Patients with Philadelphia chromosome (BCR-ABL) positive ALL
* Severe comorbidity or leukaemia-associated complications
* Known hypersensitivity to asparaginase
* History of severe pancreatitis
* History of thrombosis or pulmonary embolism
* Pre-existing clinically relevant coagulopathy
* Liver dysfunction (e.g. acute or current hepatitis, alcohol or drug abuse) or history of clinically relevant liver disease
* Bilirubin > 1.5 x Upper Limit Norm (ULN)
* Other current malignancies
* Severe psychiatric illness or other circumstances which may compromise the cooperation of the patient or the ability to give informed consent
* Body mass index > 30 kg/m²
* Known pregnancy, breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To compare the rate of patients with asparagine depletion 3 weeks after infusion of PEG-rASNase or Oncaspar® in the induction phase. | 3 weeks
  To compare the rate of patients with asparagine depletion 3 weeks after infusion of PEG-rASNase or Oncaspar® in the induction phase.

SECONDARY OUTCOMES:
Comparing of treatment arms | 62 days
  -the rate of patients with asparagine depletion
Comparing of treatment arms | 62 days
  the rate of patients with L-asparaginase (ASNase) activity levels in serum > 100 U/L
Comparing of treatment arms | 62 days
  the duration of ASNase activity levels in serum > 100 U/L and its variability pharmacokinetic parameters Cmax, t½, CLtotal, Kel, AUC0-t and AUC0-∞
Comparing of treatment arms | 62 days
  the time profiles of ASNase activity and amino acid levels Asparagine (ASN), Aspartic acid (ASP), Glutamine (GLN) and Glutamic acid (GLU) in serum
Comparing of treatment arms | 62 days
  the incidence of increased bilirubin grade III/IV
Comparing of treatment arms | 62 days
  the incidence of all other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Gökbuget, MD, Principal Investigator — Universitätsklinikum Frankfurt, Medizinische Klinik II, Theodor-Stern-Kai 7, 60590, Frankfurt
Locations (30):
- Germany (30):
  - Charité Campus Benjamin Franklin Hämatologie, Onkologie, Transfusionsmedizin Medizinische Klinik III, Berlin
  - Charité University Hospital Campus Virchow, Berlin
  - Universität Bonn, Medizinische Klinik & Poliklinik III, Bonn
  - Städtisches Klinikum Braunschweig Medizinische Klinik III, Braunschweig
  - Klinikum Carl Gustav Carus der Technischen Universität, Dresden
  - St. Johannes-Hospital, Duisburg
  - Universität Erlangen-Nürnberg Med. Klinik V/Hämatologie, Erlangen
  - Universitätsklinikum Essen Westdeutsches Tumorzentrum, Essen
  - Universitätsklinikum Frankfurt Medizinische Klinik II, Frankfurt
  - Universitätsmedizin Göttingen Hämatologie / Onkologie, Göttingen
  - Katholisches Krankenhaus Hagen gGmbH Klinik für Hämatologie und Onkologie, Hagen
  - Asklepios Klinik St. Georg Hämatologie & Stammzelltransplantation, Hamburg
  - Asklepios Klinik Altona II. Medizinische Abteilung, Hamburg
  - Evangelisches Krankenhaus Medizinische Klinik Hämatologie/Onkologie, Hamm
  - Medical University Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universität Leipzig José-Carreras-Haus Abt. Hämatologie / Onkologie, Leipzig
  - Universitätsmedizin Mainz III. Medizinische Klinik, Mainz
  - Klinikum Schwabing, Klinik für Hämatologie, Onkologie, Immunologie, Palliativmedizin, Infektiologie & Tropenmedizin, München
  - Klinikum Rechts der Isar der TU München III. Medizinische Klinik, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, 5. Medizinische Klinik, Nuremberg
  - Klinikum Oldenburg Innere Medizin II, Oldenburg
  - Klinikum Ernst von Bergmann, Zentrum für Hämatologie, Onkologie und Strahlenheilkunde, Potsdam
  - Klinikum der Universität Regensburg, Regensburg
  - Universität Rostock, Zentrum für Innere Medizin, Klinik III, Rostock
  - Robert Bosch-Krankenhaus Abt. Hämatologie / Onkologie, Stuttgart
  - Universitätsklinik Ulm Klinik für Innere Medizin III Zentrum für Innere Medizin, Ulm
  - Klinikum der Universität Würzburg, Würzburg